CLINICAL TRIAL: NCT01001741
Title: A Pilot Study of Cellular Phone Text Message Reminders to Improve HIV Medication Adherence at Independence Surgery Clinic Gaborone, Botswana
Brief Title: Pilot Study of Text Message Reminders to Improve HIV Medication Adherence in Botswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 805891; NIH: P30 AI 045008
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infections
Keywords: HIV; Antiretrovirals; Adherence; Text messaging; Antiretroviral adherence; Treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cell phone text message — We will use cellular text messages to remind patients of impending drug prescription refills and scheduled visits to their healthcare provider.

SUMMARY:
While medication adherence is critical to successful treatment of HIV, there are few studies of interventions demonstrating improvements in adherence. This may be a particular challenge in the developing world, which has a larger burden of HIV but fewer resources than industrialized countries. The investigators propose a randomized controlled trial of cellular phone text message reminders to improve medication adherence. Our pilot study will be set in a large HIV clinic in Gaborone, Botswana, where Penn researchers have collaborated on research projects in the past. The primary study outcome will be antiretroviral medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* 21 years of age or older

Exclusion Criteria:

* Subjects who do not intend to have continuous follow-up care and monthly medication refills at Independence Surgery for at least the next six months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
HIV medication adherence | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Darren Linkin, MD, Study Director — University of Pennsylvania; Harvey Friedman, MD, Principal Investigator — University of Pennsylvania; James Thompson, MBA, Study Director — Wharton Business School, UPenn; Andrew Steenhoff, Study Director — University of Pennsylvania
Locations (1):
- Independence Surgery, Gaborone, Botswana

REFERENCES:
- [Result] Reid MJ, Dhar SI, Cary M, Liang P, Thompson J, Gabaitiri L, Steele K, Mayisela S, Dickinson D, Friedman H, Linkin DR, Steenhoff AP. Opinions and attitudes of participants in a randomized controlled trial examining the efficacy of SMS reminders to enhance antiretroviral adherence: a cross-sectional survey. J Acquir Immune Defic Syndr. 2014 Feb 1;65(2):e86-8. doi: 10.1097/QAI.0b013e3182a9c72b. No abstract available. PMID 24442231
- See also: University of Pennsylvania in Botswana — http://www.uphs.upenn.edu/idd/bots.html